CLINICAL TRIAL: NCT05320991
Title: A Randomized Control Trial Employing fMRI to Investigate the Effects of Ketamine on Mentalizing and Metacognition in Healthy Volunteers
Brief Title: Effects of Ketamine on Mentalizing and Metacognition in Healthy Volunteers
Acronym: METAKETAII
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Rene Hurlemann, Professor for Psychiatry, University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: #19-03-29 (METAKETA)
Record Dates: First submitted 2022-03-14; First posted 2022-04-11 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Ketamine-Induced Psychotic Disorder; Social Cognition; Theory of Mind
Keywords: ketamine; fMRI; psychosis; mentalizing; social cognition; metacognition
MeSH Terms: conditions — Psychotic Disorders | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All investigators (except anesthesiologists) are blinded until fMRI data has been preprocessed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Participants receive a saline-solution intravenously
  Interventions: Drug: Nacl 0.9%
- Ketamine (Experimental): Participants receive ketamine (Plasma-level 100 ng/ml with an initial bolus administered as a 2 mg/ml solution)
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Ketamine is applied with a Graseby 3500 intravenous infusion pump controlled by the STANPUMP software (Steven Shafer, M.D., Anesthesiology Service, PAVAMC 3801 Miranda Ave., Palo Alto, USA). Target plasma levels are 100 ng/ml with an initial bolus administered as a 2 mg/ml solution.
  Arms: Ketamine
Drug: Nacl 0.9% — Saline solution will also be applied with the Graseby 3500 intravenous infusion pump controlled by the STANPUMP software (Steven Shafer, M.D., Anesthesiology Service, PAVAMC 3801 Miranda Ave., Palo Alto, USA).
  Arms: Placebo

SUMMARY:
Antipsychotic medication shows generally good effect sizes when looking at reduction of positive psychotic symptoms of schizophrenia, such as paranoia or delusion. However, social functioning often remains deficient in patients, meaning dopamine-receptor antagonists are not sufficient in treatment of people with schizophrenia.

A naturalistic video-based paradigm, named MASC has been used in the past to model over- and undermentalizing in patients with autism spectrum disorder and schizophrenia, since deficits in mentalizing can be explained by either overinterpreting a social situation (e.g. paranoid thoughts about intentions of others towards self) or by lacking the skill to read intentions of others.

To find out whether experimental manipulation via a non-competetive N-methyl-D-aspartate antagonist can induce difficulties with social cognition similar to those observed in people with schizophrenia, the investigators will conduct a RCT applying either ketamine or a placebo intravenously while participants are completing the above mentioned mentalizing task in the fMRI-scanner.

ELIGIBILITY:
Potential participants are excluded based on the following criteria:

* history of psychiatric/neurological disorder (self and first-degree relatives)
* learning disabilities, or loss of consciousness for more than 5 minutes
* history of alcohol or drug abuse within the last 12 months
* history of ketamine abuse
* history of complications during anesthesia (self and first-degree relatives)
* serious physical illness
* claustrophobia
* color-blindness
* metalliferous implant
* visual impairments other than corrective lenses
* injury or disease of the inner ear with loss of hearing
* consumption of any prescription or over-the-counter medication 3 days previous to the examination
* pregnancy
* currently breastfeeding a baby
* hypotension (blood pressure < 100/60)
* hypertension (blood pressure > 140/90)
* underweight (BMI <17)
* overweight (BMI ≥30)

Recruited participants are required to meet the following criteria:

* height between 150 and 195 cm
* bodyweight between 50 and 99kg
* male or female
* right-handed
* physically, neurologically and psychiatrically healthy
* non-smoker
* normal or corrected-to-normal eye-sight
* good command of German language

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2020-09-27 (Actual); Study Completion 2020-09-27 (Actual)

PRIMARY OUTCOMES:
Changes in Mentalizing/Theory of Mind | During ketamine/placebo application in MRI
  Over- and undermentalizing as characterized by the Movie for the assessment of social cognition (MASC). Higher scores on the "Mentalizing"-scale indicate better performance. Scores are divded between 4 scales (Mentalizing, No Mentalizing, Overmentalizing, Undermentalizing), each ranging from 0 to 27. Higher scores in one of the scales pertaining to "no Mentalizing, Overmentalizing or Undermentalizing mean a deficiency in mentalizing skills.
Neural response to ketamine/placebo during social cognition | During ketamine/placebo application in MRI
  fMRI imaging will be performed to measure blood oxygen level-dependent (BOLD) signal in response to mentalizing cues in the MASC-task under ketamine/placebo. BOLD-signal will be measured with T2-weighted images in a 3T MRI. Data will be analyzed using SPM 12 in MATLAB. Deviations in BOLD-activity under ketamine compared to placebo (higher or lower activity of certain voxels/clusters compared all other voxels in the brain) will mean a change in neural response due to the effect of the substance

SECONDARY OUTCOMES:
Psychotic symptom load in PANSS-Questionnaire | 10 minutes after cessation of MRI and ketamine/placebo application
  Positive and negative symptoms measured with questionnaire used in schizophrenia-research (Positive and Negative Symptom Scale). The PANSS uses a scale ranging from 1 to 7 in three different subscales (positive, 7 items; negative, 7 items; disorganized, 16 items). Higher numbers mean more psychotic symptoms.
Metacognitive-Questionnaire (MCQ) | 20 minutes after cessation of MRI and ketamine/placebo application
  Metacognitive typology as assessed with the MCQ. The MCQ is a questionnaire containing 30 items, based on a 4-point Likert scale (dont agree - strongly agree) from 1 to 4. It measures metacognitive ability in 5 subscales, each containing 6 items (Uncontrollability and Danger, Cognitive Self-Consciousness, Need to control thoughts, Positive Beliefs, Cognitive Confidence). This is a short form of the widely used Metacognitions Questionnaire that measures individual differences in a selection of metacognitive judgments and monitoring tendencies considered important in the metacognitive model of psychological disorders

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry and Psychotherapy, University Hospital Bonn, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://sites.google.com/view/bonnsocialneuroscienceunit